CLINICAL TRIAL: NCT01736332
Title: Evidence-Based Drug Policy and Legislation: Amphetamines and Opiates in Blood, Oral Fluid and Urine Following Intranasal l-Methamphetamine and Oral Poppy Seeds
Brief Title: Factors Affecting Methamphetamine and Opiates Drug Testing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 999912481; 12-DA-N481
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-03-19

CONDITIONS: Opiates; Healthy
Keywords: Methamphetamine; Amphetamines; Opiates; Oral Opiates (poppy seeds); Intranasal amphetamines

INTERVENTIONS:
Drug: Vicks VapoInhaler — 2 inhalations each nostril every 2 hours for 6 doses on day 1, one dose on morning of day 2
Other: Poppy seeds — 45 g in liquid at 9 am and 5 pm on day 1

SUMMARY:
Background:

- Some legal over-the-counter drugs (such as Vicks VapoInhaler ) and some foods (such as poppy seeds) may cause a positive screening drug test. This might look like someone used illegal drugs (such as methamphetamines or opiates) when they did not. Researchers are studying how the body handles chemicals that may test like illegal drugs and for how long they may be detected in the body. Blood, saliva, and urine samples will be collected. This study may help improve the effectiveness and accuracy of drug tests.

Objectives:

- To see how the body handles chemicals that may produce positive screening tests and how additional testing can eliminate positive drug tests from over-the-counter drugs and food.

Eligibility:

- Healthy volunteers between 18 and 65 years of age.

Design:

* Participants are screened with a physical exam, medical history, laboratory tests, and ECG.
* This study involves an overnight stay on a secure research unit and 2 days of tests.
* On the first day, participants will take Vicks VapoInhaler (two inhalations in each nostril) every 2 hours from 9 a.m. to 7 p.m. They will also take a drink containing poppy seeds twice (at about 9 a.m. and 5 p.m.).
* On the morning of the second day, participants will take the Vicks VapoInhaler just once. They will be discharged around 5 p.m.
* On both days, participants will provide blood and saliva samples several times throughout the day. All of their urine will be collected during the 2 study days....

DETAILED DESCRIPTION:
Objective: Two widely available legal products, Vicks VapoInhaler (lmethamphetamine with trace amounts of d-methamphetamine) and poppy seeds (morphine and codeine) contain small amounts of psychoactive substances that may generate positive tests for regulated drugs conducted in forensic, workplace and drug abuse treatment settings. This study evaluates the prevalence and duration of positive amphetamines and opiates drug tests in blood, oral fluid (OF) and urine.

Study population: Up to 30 healthy adults without a history of clinically significant adverse reactions to nasal or oral decongestants or stimulants, to oral opiates, or to poppy seeds, buckwheat, hazelnuts, or sesame.

Design: This is an open-label, non-treatment study in which each participant spends two days at NIDA IRP and the intervening night on the Behavioral Pharmacology Research Unit (BPRU). Vicks VapoInhaler (0.16-0.60 milligrams of l-methamphetamine and trace amounts of d-methamphetamine) is administered intranasally every two hours for six doses from 9 am to 7 pm on the first day and a seventh dose at 6 am the second day. Food grade uncooked poppy seeds (45 grams suspended in 500 milliliter of liquid) are administered orally at 9 am and 5 pm on the first day only.

Outcome measures: The primary outcome measures are prevalence of positive tests and windows of drug detection (based on concentrations in the biological matrix) of methamphetamine, l-amphetamine, morphine, and codeine in blood, OF, and urine. Secondary outcome measures are 1) performance of 2 OF collection devices (Quantisal and Oral-Eze) and an on-site OF screening test (Draeger Drug Test 5000) in comparison to liquid chromatography-tandem mass spectrometry (LCMSMS), and performance of urine screening test in comparison to gas chromatography-mass spectrometry (GC-MS). Performance parameters are prevalence of positive tests at each time point, windows of drug detection, sensitivity, and specificity for l-methamphetamine, l-amphetamine, morphine, and codeine in OF and urine. Cutoff concentrations for each matrix are those specified in the Mandatory Guidelines for Federal Workplace Drug Testing Programs; 2) detection of d-methamphetamine in any blood, OF and urine specimen; and 3) time course of these analytes in blood for comparison to other matrices, especially oral fluid/blood ratios.

Significance: These data are essential for establishing evidence-based drug policy and legislation, for establishing oral fluid drug testing by the Substance Abuse and Mental Health Services Administration, and for answering current questions about whether use of these legal products could produce positive tests in federally mandated drug testing programs.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 to 65 years.
* Able to give valid informed consent.
* Able to cooperate with all study procedures.
* Peripheral venous access adequate to allow repeated blood sampling

EXCLUSION CRITERIA:

* Current medical condition that precludes safe study participation, such as 2nd or 3rd
* Current physical dependence on any psychoactive substance other than caffeine or nicotine.

degree A-V block, acute coronary syndrome, premature atrial contractions occurring more than 3/min, or premature ventricular contractions occurring more than 1/min.

* Inability to tolerate intranasal medication administration.
* Inability to safely swallow liquids containing poppy seeds.
* History of clinically significant adverse reaction to intranasal or oral decongestants.
* History of clinically significant adverse reaction to opiates.
* History of clinically significant adverse reaction from exposure (oral, inhalational, tactile) to poppy seeds, buckwheat, hazelnuts, or sesame.
* Inability to tolerate abstinence from any medication that might adversely interact with opiates, e.g., CNS depressant, systemically acting anti-cholinergic, or monoamine oxidase inhibitor.
* Women who are pregnant or nursing.
* Use, within 7 days of initial dosing with study substances, of prescription amphetamine or opiate-like substances that are related to the substances being tested.
* Internal nasal lesions that increase risk of inhalation of Vicks VaporInhaler
* Current hypertension, cardiomyopathy,or other current medical conditions associated with increased risk from adrenergic or opioid drug administration.
* Resting blood pressure consistently >140/90 mm Hg or heart rate consistently > 90 bpm
* Resting systolic blood pressure consistently < 90
* Urine drug test positive for amphetamines or opiates
* Use of a nasal decongestant or ingested an amphetamine, opiate, CNS depressant, anticholinergic, or poppy seeds within the prior week, or a monoamine oxidase inhibitor within the prior 2 weeks
* History of psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-07-19; Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of positive tests and windows of drug detection (based on concentrations in the biological matrix) of I-methamphetamine, I-amphetamine, morphine, and codeine in blood, OF, and urine.

SECONDARY OUTCOMES:
Heart rates, blood pressure, respiratory rate | 30 hours
Performance of 2 OF collection devices (Quantisal and Oral-Eze) and an on-site OF screening test (Draeger Drug Test 5000) in comparison to LC-MS-MS and performance fo urine screening test in comparison to GC-MS. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huestis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Crivellaro M, Bonadonna P, Dama A, Senna GE, Mezzelani P, Mistrello G, Passalacqua G. Severe systemic reactions caused by poppy seed. J Investig Allergol Clin Immunol. 1999 Jan-Feb;9(1):58-9. PMID 10212860
- [Background] Dufka F, Galloway G, Baggott M, Mendelson J. The effects of inhaled L-methamphetamine on athletic performance while riding a stationary bike: a randomised placebo-controlled trial. Br J Sports Med. 2009 Oct;43(11):832-5. doi: 10.1136/bjsm.2008.048348. Epub 2008 Nov 3. PMID 18981044
- [Background] Fritschi G, Prescott WR Jr. Morphine levels in urine subsequent to poppy seed consumption. Forensic Sci Int. 1985 Feb;27(2):111-7. doi: 10.1016/0379-0738(85)90173-2. PMID 3979930